CLINICAL TRIAL: NCT05539248
Title: A Multicenter, Open-label, Multiple Ascending Dose Phase 1b/2 Trial to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of CAN106 Intravenously in Subjects With PNH Naïve to Complement-Inhibitor Treatment
Brief Title: A Study on the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of CAN106 in Subjects With PNH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CARE Pharma Shanghai Ltd. (Industry)
Responsible Party: Sponsor
Organization: CANbridge Life Sciences Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAN106-PNH-102/201; CTR20220162 (Registry Identifier: Center For Drug Evaluation, NMPA, China)
Record Dates: First submitted 2022-07-07; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-07

CONDITIONS: PNH; Hemolysis
Keywords: C5 complement inhibitor; CAN106; PNH
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation CAN106 in cohort 1 (Experimental): Subjects are administered CAN106 20 mg/kg IV maintenance dosing.
  Interventions: Drug: CAN106 20 mg/kg
- Dose escalation CAN106 in cohort 2 (Experimental): Subjects are administered CAN106 40 mg/kg IV maintenance dosing.
  Interventions: Drug: CAN106 40 mg/kg
- Dose escalation CAN106 in cohort 3 (Experimental): Subjects are administered CAN106 80 mg/kg IV maintenance dosing.
  Interventions: Drug: CAN106 80 mg/kg

INTERVENTIONS:
Drug: CAN106 20 mg/kg — Induction and maintenance dosing for cohort 1:
  12 mg/kg on Day 1, 16 mg/kg on Day 8, and 20 mg/kg on Day 15 and every 4 weeks thereafter;
  Arms: Dose escalation CAN106 in cohort 1
Drug: CAN106 40 mg/kg — Induction and maintenance dosing for cohort 2:
  30 mg/kg on Day 1, and 40mg/kg on Day 8 and every 4 weeks thereafter；
  Arms: Dose escalation CAN106 in cohort 2
Drug: CAN106 80 mg/kg — Induction and maintenance dosing for cohort 3:
  60 mg/kg on day 1, and 80 mg/kg on day 15 and every 8 weeks thereafter.
  Arms: Dose escalation CAN106 in cohort 3

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, efficacy, pharmacokinetics, and pharmacodynamics of CAN106 administered intravenously to subjects with PNH who have not previously been treated with a complement inhibitor.

DETAILED DESCRIPTION:
This is an open-label, multiple dose escalation study to assess the safety, tolerability, efficacy, PK, PD and immunogenicity of CAN106 given as an IV infusion. The data presented is up to the primary completion date of the study and is for the 26-week primary evaluation period. The study also includes an extension period of up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age.
2. Body weight ≥40 kg at screening.
3. Documented diagnosis of PNH within 6 months prior to screening, confirmed by high-sensitivity flow cytometry evaluation of red blood cells (RBCs), with granulocyte or monocyte clone size of ≥10%.
4. LDH level ≥ 1.5 X ULN at screening.
5. Mean hemoglobin(Hb)<10 g/dL for those who have not received blood. transfusion at screening, based on 2 measurements from separate blood samples collected at interval of 2-8 weeks apart prior to the first dosing. Or hemoglobin < 10 g/dL at the first screening and then with subsequent red blood cell transfusions.
6. Presence of 1 or more of the following PNH-related signs or symptoms within 3 months of Screening: fatigue, hemoglobinuria, abdominal pain, shortness of breath (dyspnea), anemia (hemoglobin < 10 g/dL), history of a major adverse vascular event (including thrombosis), dysphagia, or erectile dysfunction; or history of pRBC transfusion due to PNH.
7. All patients must be vaccinated against meningococcal infections within 3 years prior to, or at the time of, initiating study drug. Patients who initiate study drug treatment less than 2 weeks after receiving a meningococcal vaccine must receive treatment with appropriate prophylactic antibiotics until 2 weeks after vaccination.
8. If available, Haemophilus influenzae type b and Streptococcus pneumoniae vaccines can be administered according to national vaccine guidelines, and antibiotic prophylaxis should be given until 2 weeks after vaccination if the vaccines are administered within 14 days prior to administration.
9. All females of childbearing potential and all males must be willing to use at least one highly effective method of contraception from signing of informed consent until 8 months after the last dose of CAN106 Injection; Male subjects with female partners of childbearing potential must be willing to use condoms in addition to using a highly effective method of contraception.
10. Subjects should be willing to sign the informed consent forms and comply with the study visit.

Exclusion Criteria:

1. Current or previous treatment with a complement inhibitor.
2. Positive pregnancy test on day 1, or female patients who are planning to become pregnant or are pregnant or breastfeeding.
3. Participation in an interventional clinical study within 28 days before initiation of dosing on Day 1, or within 5 half-lives of the investigational product, whichever is greater.
4. Platelet count < 30 × 10^9/L at Screening.
5. Absolute neutrophil count < 0.5 × 10^9/L at Screening.
6. Alanine aminotransferase (ALT) > 3 × ULN, or both direct bilirubin and alkaline phosphatase (ALP) > 2 × ULN during the screening period.
7. Serum creatinine > 2.5 × ULN and creatinine clearance < 30 mL/min as calculated by the Cockcroft-Gault formula during the screening period.
8. History of malignancy within 5 years of Screening with the exception of nonmelanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
9. History of bone marrow transplantation.
10. Major surgery within 90 days prior to screening.
11. History of N. meningitidis infection or unexplained, recurrent infection.
12. Known or suspected hereditary complement deficiency.
13. Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing
14. Presence of fever ≥38°C within 7 days prior to study drug administration.
15. Having received splenectomy within 6 months prior to screening.
16. Known history of severe allergic or anaphylactic reactions to antibiotics and are unwilling to use prophylaxis as specified in the protocol.
17. Patients are excluded if they are taking any of the following medications and are not on a stable regimen(as judged by investigator) for the time period indicated prior to screening:

    1. Erythropoietin or immunosuppressants for at least 8 weeks;
    2. Corticosteroids for at least 4 weeks;
    3. Vitamin K antagonists with a stable international normalized ratio for 4 weeks;
    4. Iron supplements or folic acid for at least 4 weeks;
    5. Low molecular weight heparin for at least 4 weeks.
18. Known allergy to excipients of CAN106 or allergy to Chinese hamster ovary cell proteins.
19. Immunization with a live-attenuated vaccine 1 month prior to dosing on day 1.
20. Known or suspected history of drug or alcohol abuse or dependence within 1 year prior to the start of Screening.
21. Inability to comply with study requirements.
22. History of or ongoing major cardiac, pulmonary, renal, endocrine, or hepatic disease (eg, active hepatitis) that, in the opinion of the Investigator or Sponsor, precludes the patient's participation in an investigational clinical trial.
23. Known medical or psychological condition(s) or risk factor that, in the opinion of the Investigator, might interfere with the patient's full participation in the study, pose any additional risk for the patient, or confound the assessment of the patient or outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) of multiple doses of CAN106 as assessed by CTCAE v5.(Phase 1b) | 182 days
  TEAEs were defined as adverse events (AE) that occurred after dosing on Day 1 and up to 28 days after the last dose of CAN106, include adverse events (AEs), serious adverse events (SAEs), AEs of special interest (AESIs), abnormal laboratory data compared with baseline, vital signs, and electrocardiograms (ECGs)
Percent Change In Lactate Dehydrogenase (LDH) Levels Normalization From Baseline to Day 182(Phase 2) | Baseline, Day 182
  Baseline is defined as the average of all available assessments prior to first CAN106 infusion.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) - Pharmacokinetics parameter | 182 days
  Area under the plasma concentration versus time curve to the last visit (AUC)
Maximum Plasma Concentration (Cmax) - Pharmacokinetics parameter | 182 days
  Peak plasma concentration
Time to Maximum Concentration (Tmax) - Pharmacokinetics parameter | 182 days
  Time to reach maximum of concentration (days)
t1/2 - Pharmacokinetics parameter | 182 days
  Terminal elimination half-life
PD parameters-free C5 | 182 days
  Maximal change from baseline in free C5 concentrations at each of scheduled post baseline assessment time-points (µg/ml)
PD parameters-CH50 | 182 days
  Maximal change from baseline total complement activity (CH50) at each of scheduled post baseline assessment time-points (%)
PD parameters- total C5 | 182 days
  Measure the absolute change from baseline in total C5 concentrations at each of scheduled post baseline assessment time-points (µg/ml)
Immunogenicity | 182 days
  Anti-drug Antibody (ADA) titers
Changes from Baseline in Serum Lactate Dehydrogenase (LDH) Level | 182 days
  Changes from baseline in serum LDH level to Day 182
Percent Change In Free Hemoglobin Level From Baseline to Day 182 | 182 days
  Changes from baseline in free hemoglobin level at each of the scheduled post-baseline time-points
Percent Change In Haptoglobin Levels From Baseline to Day 182 | 182 days
  Changes in haptoglobin from baseline to each of the scheduled post-baseline time-points
Changes in scores of patient-reported outcomes as measured by FACIT-Fatigue from Baseline to Day 182 | 182 days
  The FACIT-F is a 13-item, self-reported PRO measure assessing an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related QoL in patients with cancer and other chronic illnesses. The FACIT-fatigue assesses the level of fatigue using a 4-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating greater fatigue
Changes in scores of patient-reported outcomes as measured by European Organization for Research and Treatment of Cancer [EORTC]- Quality of life questionnaire-core 30 (QLQ-30) | 182 days
  EORTC QLQ-C30 is a self-reported, 30-item generic questionnaire developed to assess 15 domains: global health status scale, five functional scales (physical, role, emotional, cognitive, and social functioning) and nine symptom scales (fatigue, nausea, vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). All the scales range from 0 to 100. A high score on the functional scales represents a high level of functioning, and a high score on the symptom scales represents a high level of symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, MD, Principal Investigator — Peking Union Medical College Hospital; Hongzhong Liu, MMed, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China